CLINICAL TRIAL: NCT06630585
Title: GIP/GLP-1RA as Adjunctive to Automated Insulin Delivery in Adults With Type 1 Diabetes: A Prospective, Randomized, Clinical Study - The AID-JUNCT Trial
Brief Title: GIP/GLP-1RA as Adjunctive to Automated Insulin Delivery in Adults With Type 1 Diabetes
Acronym: AID-JUNCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Kantonsspital Olten (Other); Luzerner Kantonsspital (Other); Clinique des Grangettes, Chêne-Bougeries (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01947
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 diabetes; Adjuvant therapy; Incretins; GIP/GLP-1RA
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Participants in this arm will use their standard of care (SoC)
- Standard of Care + Drug (Experimental): Participants in this arm will use their standard of care (SoC) plus tirzepatide (titrated to reach a minimum accepted dose.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide is a clear, colorless to slightly yellow solution available in cartons containing four pre-filled single-dose pens or one single-dose vial: 2.5 mg, 5 mg, 7.5 mg, 10 mg, 12.5 mg, or 15 mg per 0.5 mL in a single-dose pen or vial.
  In this study, the investigators will start with the recommended starting dosage of tirzepatide: 2.5 mg injected subcutaneously once weekly (for four weeks). After four weeks, the dosage will be increased to 5 mg once weekly injected subcutaneously for 12 weeks.
  Other Names: GIP/GLP-1RA
  Arms: Standard of Care + Drug

SUMMARY:
Blood glucose management in type 1 diabetes (T1D) remains a challenge, with only ~30% of adults within the recommended consensus guidelines. Novel drugs like glucagon-like peptide-1 receptor agonists (GLP-1RAs) and glucose-dependent insulinotropic polypeptide (GIP)/GLP-1RAs have emerged as promising add-ons to insulin in T1D.

This application has been designed to test in a prospective study whether adding a new medicine called tirzepatide (GIP/GLP-1RA) to the usual insulin therapy would make a difference for people with T1D in terms of better glucose control.

DETAILED DESCRIPTION:
Glycemic control in type 1 diabetes (T1D) remains a challenge, with ~30% of adults achieving an A1c target of 7%. The glucagon-like peptide-1 receptor agonists (GLP-1RAs) and glucose-dependent insulinotropic polypeptide (GIP)/GLP-1RAs have emerged as a promising therapy in T1D. Retrospective studies have shown patients with T1D can significantly improve glycemic control with a reduction in insulin dose and body weight when long-acting GLP-1RAs or GIP/GLP-1RAs are added to insulin therapy. However, randomized controlled trials (RCT) are still lacking.

This is a prospective, randomized, open-label design. The investigators will enroll 42 participants over 18 years of age with confirmed T1D diagnosis ≥6 months, currently on automatic insulin delivery (AID) therapy for at least three months, with A1C ≥6.5% and ≤10%and BMI ≥23 kg/m2. Participants will be randomized in a 1:1 ratio to either tirzepatide 5.0 mg or continue with the Standard of Care (SoC) for 12 weeks (after a titration phase with the lowest dose of 2.5 mg). The primary endpoint is continuous glucose monitoring (CGM) percent time spent between 3.9 and 10.0 mmol/L (TIR) from baseline to follow-up after 12 weeks of treatment. Secondary endpoints include the change in 24/7 CGM percent time >10.0 mmol/L, 24/7 CGM percent time >13.9 mmol/L, 24/7 CGM percent time <3.9 mmol/L, 24/7 CGM percent time <3.0 mmol/L and the change in body mass index (BMI).

This is the first prospective study to investigate the efficacy and safety of tirzepatide (GIP/GLP1-RAs) as an adjuvant therapy to AID. This study may contribute unique data to significantly improving glucose outcomes, reducing the T1D burden, improving the quality of life, and re-directing attention to further treatment in T1D beyond insulin therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with diagnosed T1D for at least 12 months.
2. Aged between 18 to 65 years old (inclusive).
3. Currently on AID therapy for at least three months.
4. HbA1C higher or equal to 6.5% and less or equal to 10%.
5. BMI ≥23 kg/m2.
6. Willing to use once-weekly tirzepatide for at least 16 weeks (including four weeks of up-titration and 12 weeks of treatment)
7. Willing to wear a Dexcom G7 Sensor and share devices (AID) data uploads.
8. Willingness not to start any new non-insulin glucose-lowering agent during the trial (including metformin/biguanides, pramlintide, DPP-4 inhibitors, sodium-glucose cotransporter 2 inhibitors [SGLT2 inhibitors], and nutraceuticals).
9. A stable weight (± 5%) in the last 90 days or more before the screening and agree to not initiate a diet and/or exercise program during the study to reduce body weight other than the lifestyle and dietary measures for diabetes treatment.
10. Females with childbearing potential and males (if apply) must be willing to use reliable contraceptive methods (for the contraceptives study guidelines. See Annex 7 of the protocol)
11. An understanding and willingness to follow the protocol and signed informed consent.

Exclusion Criteria:

1. History of diabetic ketoacidosis requiring hospitalization in the past six months.
2. History of severe hypoglycemic event (Level 3, defined as seizure or loss of consciousness) in the past six months.
3. Uncontrolled Diabetic retinopathy or maculopathy
4. Severe gastroparesis.
5. Less than 12 months of insulin treatment.
6. Estimated glomerular filtration rate (eGFR) lab value below 30 mL/min/1.73 m2 by the CKD-EPI formula(99).
7. Pregnancy or intention to become pregnant during the trial (See annex 7).
8. Currently breastfeeding or planning to breastfeed.
9. Currently uncontrolled seizure disorder.
10. History of allergy to GIP/GLP-1RAs or its excipients.
11. Personal or family history of multiple endocrine neoplasia type 2 (MEN-2) or medullary thyroid carcinoma.
12. Screening calcitonin above or equal to 35 ng/L.
13. Planned any surgery during the study duration.
14. Have uncontrolled hypertension (systolic BP above or equal to 160 mmHg and/or diastolic BP above or equal to 100 mmHg). If a participant is on anti-hypertensive therapies, doses must be stable for 30 days before screening. For participants with uncontrolled hypertension at the screening visit, antihypertensive medication may be started or adjusted.
15. Personal history of one of the following cardiovascular conditions (within two months before the screening): acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, or hospitalization due to congestive heart failure (CHF).
16. Conditions that may increase the risk of induced hypoglycemia, such as CHF with NYHA Functional Classification III or IV or adrenal insufficiency.
17. Have a history of documented human immunodeficiency virus (HIV) infection.
18. Have an uncontrolled cardiac arrhythmia based on an electrocardiogram (ECG) at the screening time and the investigator's discretion.
19. Cystic fibrosis.
20. Patient with a history of gastric bypass (bariatric) surgery, sleeve gastrectomy, or restrictive bariatric surgery, such as Lap-Band® or gastric banding.
21. Uncontrolled thyroid disease as judged by the investigator
22. Serum triglycerides higher than 5.7 mmol/L (500 mg/dL) at the screening. If a participant is on lipid-lowering therapies, doses must be stable for 30 days before screening.
23. Personal history of acute or chronic pancreatitis. A participant with a history of acute pancreatitis caused by gallstones may be included in the study if the participant has had a cholecystectomy to resolve the problem.
24. Acute or chronic hepatitis other than MASLD.
25. Have a history of symptomatic gallbladder disease within the past two years (unless the participant has had a cholecystectomy to resolve the problem).
26. History of malignancy requiring chemotherapy, surgery, or radiation (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) in the previous five years.
27. Active or unstable major depressive disorder (MDD) or other severe psychiatric disorder (such as known drug or alcohol abuse, diagnosed eating disorder, or any other uncontrolled psychiatric disorder) that, in the investigator's opinion, may preclude the participant from following and completing the protocol.
28. Treatment with non-insulin glucose-lowering agents other than metformin (on a stable dose 30 days before the study)
29. Weight loss medications in the past three months.
30. Participants who are anticipated to receive, are receiving, or have received within three months before the screening (more than two weeks and more or equal to 10mg prednisolone-equivalent) chronic systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, single intraarticular injection, or inhaled preparations).
31. Have current treatment with (or history of, within three months before screening) medications that may significantly affect glucose metabolism.
32. Use of investigational drugs within five half-lives before screening.
33. Participation in another study with an investigational drug within the 30 days preceding and during the present study.
34. Current enrollment in another clinical trial unless approved by the investigator of both studies and if the clinical trial is a non-interventional registry trial.
35. Have evidence of a significant active, uncontrolled medical condition or a history of any medical problem capable of constituting a risk when using the study devices or interfering with following study procedures or the interpretation of data, as judged by the study physician at screening.
36. The enrolment of the investigator, his/her family members, employees, and other dependent persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change TIR | At week 16 of treatment.
  Mean difference in 24/7 CGM percentage time spent between 3.9 and 10 mmol/L (TIR) between groups.

SECONDARY OUTCOMES:
Glycated Hemoglobin | At week 16 of treatment.
  Mean difference between groups Glycated Hemoglobin.
CGM-measured TIR between 0700 and 2300 (TIR7-23) | At week 16 of treatment.
  Mean difference between groups in CGM-measured TIR between 0700 and 2300 (TIR7-23).
CGM-measured time in the tight range (TTR, 3.9-7.8 mmol/L) | At week 16 of treatment.
  Mean difference between groups in CGM-measured time in the tight range (TTR, 3.9-7.8 mmol/L).
24/7 CGM-measured percent time >10.0 mmol/L | At week 16 of treatment.
  Mean difference between groups in 24/7 CGM-measured percent time >10.0 mmol/L
24/7 CGM-measured percent time >13.9 mmol/L | At week 16 of treatment.
  Mean difference between groups in 24/7 CGM-measured percent time >13.9 mmol/L
24/7 CGM-measured percent time <3.9 mmol/L | at week 16 of treatment
  Mean difference between groups in 24/7 CGM-measured percent time <3.9 mmol/L
24/7 CGM-measured percent time <3.0 mmol/L | At week 16 of treatment.
  Mean difference between groups in 24/7 CGM-measured percent time <3.0 mmol/L
24/7 Total Daily Insulin (TDI) | At week 16 of treatment.
  Mean difference between in 24/7 Total Daily Insulin (TDI)

OTHER OUTCOMES:
CGM-measured TIR between 0700 and 2300 (TIR7-23) | At week 8, 12 and 16 of treatment.
  Mean difference between groups in CGM-measured TIR between 0700 and 2300 (TIR7-23).
24/7 CGM-measured percent time >10.0 mmol/L | At week 8, 12 and 16 of treatment.
  Mean difference between groups in 24/7 CGM-measured percent time >10.0 mmol/L
24/7 CGM-measured percent time >13.9 mmol/L | At week 8, 12 and 16 of treatment.
  Mean difference between groups in 24/7 CGM-measured percent time >13.9 mmol/L
24/7 CGM-measured percent time <3.9 mmol/L | At week 8, 12 and 16 of treatment.
  Mean difference between groups in 24/7 CGM-measured percent time <3.9 mmol/L
24/7 CGM-measured percent time <3.0 mmol/L | At week 8, 12 and 16 of treatment.
  Mean difference between groups in 24/7 CGM-measured percent time <3.0 mmol/L
CGM-measured glucose variability (CV) | At week 8, 12 and 16 of treatment.
  CGM-measured glucose variability measured with the coefficient of variation (CV)
24/7 Total Daily Insulin (TDI) | At week 8, 12 and 16 of treatment.
  Mean difference between in 24/7 Total Daily Insulin (TDI)
24/7 Total Daily Bolus (TDBo) | At week 8, 12 and 16 of treatment.
  Mean difference between in 24/7 Total Daily Bolus (TDBo)
Body Weight (BW) | At week 16 of treatment.
  Mean difference between groups in BW
Waist Circumference (WC) | At week 16 of treatment
  Mean difference between groups in WC
Hip circumference | At week 16 of treatment.
  Mean difference between the groups in hip circumference
Waist-to-hip ratio | At week 16 of treatment.
  Mean difference between groups in Waist-to-hip ratio
% Fat mass | At week 16 of treatment.
  Mean difference between groups in % fat mass
Fat mass index | At week 16 of treatment.
  Mean difference between groups in Fat mass index
Visceral adipose tissue | At week 16 of treatment.
  Mean difference between groups in visceral adipose tissue
Lean Mass Index | At week 16 of treatment.
  Mean difference between groups in Lean Mass Index
Appendicular Lean Mass Index | At week 16 of treatment.
  Mean difference between groups in Appendicular Lean Mass Index
Cholesterol LDL | At week 16 of treatment.
  Mean difference between groups in Cholesterol LDL
Cholesterol HDL | At week 16 of treatment.
  Mean difference between groups in Cholesterol HDL
Cholesterol non-HDL | At week 16 of treatment.
  Mean difference between groups in cholesterol non-HDL
Triglycerides | At week 16 of treatment.
  Mean difference between groups in Triglycerides
TG-glucose index | At week 16 of treatment.
  Mean difference between groups in TG-glucose index
Systolic blood pressure | At week 16 of treatment.
  Mean difference between groups in systolic blood pressure
Diastolic blood pressure | At week 16 of treatment.
  Mean difference between groups in diastolic blood pressure
Albumin to Creatinine Ratio | At week 16 of treatment.
  Mean difference between groups in Albumin to Creatinine Ratio
Hepatic Steatosis Index (HSI) | At week 16 of treatment.
  Mean difference between groups in HSI
Fibrosis Score (FIB-4) | At week 16 of treatment.
  Mean difference between groups in FIB-4

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zueger, PD Dr. med., Principal Investigator — Kantonsspital Olten
Locations (3):
- Switzerland (3):
  - DiaCenTRE - Hirslanden Clinique des Grangettes, Chêne-Bougeries, Canton of Geneva
  - Kantonsspital Olten, Olten, Canton of Solothurn
  - Luzerner Kantonspital, Lucerne

IPD SHARING:
Plan to Share IPD: No